CLINICAL TRIAL: NCT03316560
Title: A Phase 1/2 Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of AGTC-501 (rAAV2tYF-GRK1-RPGR) and a Phase 2 Randomized, Controlled, Masked, Multi-center Study Comparing Two Doses of AGTC-501 in Male Subjects With X-linked Retinitis Pigmentosa Confirmed by a Pathogenic Variant in the RPGR Gene
Brief Title: Safety and Efficacy of rAAV2tYF-GRK1-RPGR in Subjects With X-linked Retinitis Pigmentosa Caused by RPGR Mutations
Acronym: HORIZON
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-RPGR-001 HORIZON
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; retinal degeneration; RPGR; adeno-associated virus; gene therapy; AAV
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Phase 1/2 Dose Escalation (Experimental): Male subjects at least 18 y/o treated with Dose 1 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- Group 2: Phase 1/2 Dose Escalation (Experimental): Male subjects at least 18 y/o treated with Dose 2 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- Group 3 Phase 1/2 Dose Escalation (Experimental): Group 3 male subjects at least 18 y/o treated with Dose 3 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- Group 4 Phase 1/2 Dose Escalation (Experimental): Group 4 male subjects at least 6 y/o treated with Dose 3 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- Group 5 Phase 1/2 Dose Escalation (Experimental): Male subjects at least 18 y/o treated with Dose 5 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- Group 6 Phase 1/2 Dose Escalation (Experimental): Male subjects at least 18 y/o treated with Dose 6 of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR

INTERVENTIONS:
Biological: rAAV2tYF-GRK1-RPGR — Adeno-associated virus vector expressing a human RPGR gene

SUMMARY:
This study will evaluate the safety and efficacy of a recombinant adeno-associated virus vector (rAAV2tYF-GRK1-RPGR) in patients with X-linked retinitis pigmentosa caused by RPGR mutations.

DETAILED DESCRIPTION:
This protocol includes a non-randomized, open-label, Phase 1/2 study (HORIZON). Approximately 30 participants will be enrolled into the dose escalation study (HORIZON). Each participant will receive the study agent by subretinal injection in one eye on a single occasion. Enrollment will begin with the lowest dose and will proceed to higher doses only after review of safety data by a Data and Safety Monitoring Committee (DSMC). There are a total of 15 visits over approximately 36 months, and long-term follow-up evaluations annually at years 4 and 5.

ELIGIBILITY:
Phase 1/2 Dose Escalation Inclusion Criteria:

* Male subjects with a documented RPGR mutation
* Clinical diagnosis of X-linked retinitis pigmentosa (XLRP)
* Best-corrected visual acuity not better than 78 ETDRS letters (20/32) in the study eye;
* Ability to perform tests of visual and retinal function and structure and ability to comply with other research procedures;
* Detectable baseline mean macular sensitivity, as measured by microperimetry.
* Have detectable Ellipsoid Zone (EZ) line during the pre-treatment period as assessed by OCT and confirmed by the CRC.

Phase 1/2 Dose Escalation Exclusion Criteria:

* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints or increase the risk of surgical complications (for example, glaucoma, corneal or lenticular opacities, diabetic retinopathy, retinal vasculitis);
* Use of anti-coagulant agents that may alter coagulation within 7 days prior to study agent administration;
* Use of systemic corticosteroids or other immunosuppressive medications within 3 months prior to enrollment;
* Any other condition that would prevent a subject from completing follow-up examinations during the course of the study;
* Any other condition or reason that, in the opinion of the investigator, makes the subject unsuitable for the study;
* Previous receipt of any AAV gene therapy product;
* Monocular or having BCVA less than 20/800 in the fellow eye

Ages: 6 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of Adverse Events | Day 0 - Month 36
  Number and proportion of participants experiencing Grade 3 or higher local (ocular) or systemic treatment-emergent adverse events that occur during the 36 months after study agent administration; number and proportion of participants experiencing treatment-emergent AEs, including treatment-emergent serious AEs;
Number and proportion of participants experiencing abnormal clinically relevant hematology or clinical chemistry parameters. | Day 0 - Month 36

SECONDARY OUTCOMES:
Changes from baseline in visual function as measured by mesopic microperimetry in the treated eye compared to the untreated eye | Day 0 - Month 36
Changes from baseline in visual acuity | Day 0 - Month 36
Changes from baseline in retinal structure as assessed by spectral-domain optical coherence tomography (SD-OCT) | Day 0 - Month 36
Changes from baseline in quality of life questionnaire responses | Day 0 - Month 36
Change from baseline in visual function by light-adapted perimetry | Day 0 - Month 36
Change from baseline in fundus imaging | Day 0 - Month 36
Change from baseline in full-field light sensitivity threshold (FST) | Day 0 - Month 36
Changes from baseline in visual function by dark-adapted full field perimetry (for subjects treated peripherally) | Day 0 - Month 36

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Duke University, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876
- [Derived] Alibhai AY, De Pretto LR, Yaghy A, Woo KM, Dos Santos Xilau NR, Siddiqui H, Pandiscio CA, Homer A, Curtiss D, Waheed NK. Comparing the Thin Plate Spline and Gaussian Interpolation Methods in Generating Hill of Visions for X-Linked Retinitis Pigmentosa Patients. Transl Vis Sci Technol. 2024 Dec 2;13(12):26. doi: 10.1167/tvst.13.12.26. PMID 39680391